CLINICAL TRIAL: NCT05389514
Title: Intermediate-size Patient Population IND for Treatment of KRAS G12V-mutant Tumors With Gene-engineered KRAS G12V-reactive T Cells
Brief Title: Intermediate-size IND for Treatment of KRAS G12V-mutant Tumors
Status: Temporarily not available | Type: Expanded Access
Sponsor: Providence Health & Services (Other)
Responsible Party: Sponsor
Other Study IDs: 2020000471
Record Dates: First submitted 2022-05-19; First posted 2022-05-25 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: KRAS G12V Mutant Advanced Epithelial Cancers
MeSH Terms: interventions — Cyclophosphamide; Gemcitabine; pembrolizumab; Insulin Infusion Systems

STUDY DESIGN:
Expanded Access Types: Intermediate, Treatment

INTERVENTIONS:
Drug: Cyclophosphamide — Patients will receive a single dose of cyclophosphamide 60 mg/kg IV in 250 ml D5W over 2 hours on Day -3.
  Other Names: Cytoxan; Cytoxan Lyophilized; Cy
Drug: Gemcitabine — Patients will receive a single dose of gemcitabine 600 mg/mg2 IVPB over 30 minutes on Day -2.
  Other Names: Gemzar
Drug: Pembrolizumab — Patients will receive the anti-PD-1 immune checkpoint inhibitor pembrolizumab 200 mg IV over 30 minutes on Day -1 and will be dosed every 3 weeks.
  Other Names: KEYTRUDA; MK-3475
Biological: Cell Infusion — Patient's T cells will be administered at a dose of between 1 x 10^9 to 5.0 x 10^10 TCR-transduced lymphocytes, which is a dose of genetically modified T cells that can be safely administered and is capable of mediating tumor regression in some patients with metastatic cancers.
  The cells are to be infused intravenously over approximately 30 minutes via non-filtered tubing, gently agitating the bag during infusion to prevent cell clumping.

SUMMARY:
This intermediate-size IND will treat participants with incurable, advanced or metastatic cancer, harboring KRAS G12V mutation and appropriate HLA class II match (HLA-DRB1*07:01).

DETAILED DESCRIPTION:
This study will treat two identified patients with metastatic pancreatic adenocarcinoma and metastatic pancreatic cancer who have both been treated with standard of care therapies and found to have disease progression. Both of these patients have KRAS G12V mutations in their cancers and express the HLA-DRB1*07:01 HLA class II molecule. As such, they are candidates for adoptive cell therapy with autologous gene-engineered T cells expressing HLA-DRB1*07:01-restricted KRAS G12V reactive T-cell receptors (TCR).

Adoptive T-cell therapy is a type of immunotherapy which involves isolation of T cells from a patient, followed by an amplification of those T cells in the lab to large numbers, and reinfusion of the T cells back to the patient.

In addition to the two identified patients, the protocol will remain open for additional participants with incurable, advanced or metastatic cancer, harboring KRAS G12V mutation, and appropriate HLA class II match (DRB1*07:01).

ELIGIBILITY:
Patients with incurable, advanced or metastatic cancer, harboring KRAS G12V mutation, and appropriate HLA class II match (HLA-DRB1*07:01)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Taylor, MD, Principal Investigator — Providence Health & Services